CLINICAL TRIAL: NCT06609577
Title: Personalized Ultrasound Guided Pacing of the External Diaphragm to Improve Outcomes in Patients Undergoing Invasive Mechanical Ventilation: a Randomized Controlled Trial
Brief Title: Personalized Ultrasound-Guided External Diaphragm Pacing to Improve Outcomes in Invasive Mechanically Ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daishan Jiang (Other)
Responsible Party: Sponsor-Investigator, Daishan Jiang, Senior Attending Physician, Affiliated Hospital of Nantong University
Organization: Affiliated Hospital of Nantong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-L146
Record Dates: First submitted 2024-09-17; First posted 2024-09-24 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Failure; Mechanical Ventilation
Keywords: External Diaphragm Pacing; Diaphragm Ultrasound; Mechanical Ventilation; Ventilator Weaning; Critical Care
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Control group (No Intervention): Received standard mechanical ventilation withdrawal protocol without diaphragmatic external pacing
- Invention group (Experimental): Diaphragm function was monitored by diaphragmatic ultrasound to personalize the intensity of diaphragm extracorporeal pacing.
  Interventions: Device: Diaphragm Ultrasound-Guided External Diaphragm Pacing

INTERVENTIONS:
Device: Diaphragm Ultrasound-Guided External Diaphragm Pacing — This intervention, Diaphragm Ultrasound-Guided External Diaphragm Pacing (DU-EDP), is distinguished by its personalized approach, where diaphragm pacing is dynamically adjusted based on real-time diaphragm function measurements obtained through bedside diaphragm ultrasound (DU). Unlike standard external diaphragm pacing (EDP) interventions that use uniform pacing parameters, DU-EDP allows for the customization of pacing intensity, frequency, and duration for each patient. This intervention specifically integrates novel diaphragm function indices, such as diaphragm thickening fraction (DTF) and diaphragmatic rapid shallow breathing index (D-RSBI), to enhance precision in weaning from mechanical ventilation. The combination of these advanced metrics with real-time ultrasound guidance makes DU-EDP a highly individualized and innovative intervention for critically ill, mechanically ventilated patients.
  Arms: Invention group

SUMMARY:
This study aims to explore whether personalized external diaphragm pacing (EDP) guided by real-time diaphragm ultrasound (DU) can improve outcomes for patients on invasive mechanical ventilation. Diaphragm ultrasound will be used to assess each patient's diaphragm function and adjust the pacing intensity, creating a customized treatment plan. By using this individualized approach, the investigators hope to prevent diaphragm muscle weakening, which is a common issue during prolonged ventilation, and improve the chances of successful weaning from the ventilator. The study will also incorporate advanced diaphragm function metrics, such as diaphragm thickening fraction (DTF) and diaphragmatic rapid shallow breathing index (D-RSBI), to enhance the accuracy of treatment and improve patient recovery. This trial aims to improve overall outcomes and quality of care for patients requiring long-term mechanical ventilation.

DETAILED DESCRIPTION:
This study investigates the efficacy of a personalized external diaphragm pacing (EDP) protocol, dynamically guided by diaphragm ultrasound (DU), in improving outcomes in mechanically ventilated patients. Unlike traditional EDP systems that use uniform pacing parameters, this study introduces an individualized approach that uses diaphragm function-monitored by real-time DU-to adjust pacing intensity, frequency, and duration for each patient. The goal is to optimize diaphragm activity, prevent muscle atrophy, and increase the likelihood of successful weaning from mechanical ventilation.

Key innovations in this study include the integration of novel diaphragmatic performance indicators such as diaphragmatic thickening fraction (DTF) and diaphragmatic rapid shallow breathing index (D-RSBI). These parameters will be used to assess diaphragm function more accurately than conventional methods and to inform adjustments to the stimulation regimen. By targeting ventilator-induced diaphragm dysfunction (VIDD) and preventing muscle weakness, this personalized approach aims to improve clinical outcomes, reduce ventilation time and facilitate recovery in critically ill patients.

The study will be a randomized controlled design comparing the effectiveness of personalized ultrasound-guided EDP to standard mechanical ventilation weaning protocols. Participants will be critically ill, mechanically ventilated patients requiring long-term respiratory support. Outcomes will include weaning success rate, time on mechanical ventilation, and overall patient survival and recovery rates. The trial aims to advance critical care protocols by integrating personalized technology to improve patient outcomes in the mechanical ventilation setting.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age undergoing invasive mechanical ventilation.
2. Expected duration of mechanical ventilation ≥48 hours.

Exclusion Criteria:

1. ICU expected length of stay less than 48 hours
2. severe phrenic nerve or diaphragmatic injury that is unable to respond to diaphragmatic pacing.
3. Patients who have received or are scheduled to receive other respiratory assistance or diaphragmatic pacing interventions.
4. Patients with end-stage disease with an expected survival of &amp;lt;6 months.
5. Patients who are unable to be weaned from mechanical ventilation, such as patients with severe brain injury or paraplegia.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Weaning Success Rate | Assessed 48 hours and 72 hours after weaning to ensure no need for reintubation or mechanical support.
  The proportion of patients who are successfully weaned off mechanical ventilation for at least 48 hours without respiratory failure or reintubation.

SECONDARY OUTCOMES:
Total Duration of Invasive Mechanical Ventilation | From the date of randomization until the time of successful weaning or patient discharge, whichever comes first, assessed up to 90 days after admission.
  The total duration of invasive mechanical ventilation, measured in hours, from the initiation of mechanical ventilation post-randomization until successful weaning, defined as 48 consecutive hours of spontaneous breathing without any invasive mechanical ventilation support.
ICU Length of Stay | From the date of randomization until the date of ICU discharge, assessed up to 90 days after admission..
  The total number of days the patient stays in the Intensive Care Unit (ICU), from the date of ICU admission until the date of ICU discharge.
30-Day and 90-Day Survival Rates | Follow-up conducted at 30 days and 90 days after admission
  The survival rates of patients at 30 and 90 days after successful weaning, assessing outcomes.
Prevention of Diaphragm Atrophy | From the date of randomization, assessed at baseline (within 24 hours post-randomization), on days 3 during treatment, and at the time of successful weaning, or until the date of patient discharge, , whichever comes first, assessed up to 90 days.
  Changes in diaphragm thickness and prevention of muscle atrophy, assessed by ultrasound, comparing baseline values (at randomization) with measurements taken during treatment and at follow-up intervals. Measurements will be performed at predefined time points to evaluate the impact of treatment on diaphragm preservation.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No